CLINICAL TRIAL: NCT06988748
Title: The Effect of Tonsillectomy Diet Education on Bleeding and Pain After Adenotonsillectomy in Children
Brief Title: Diet Education and Postoperative Outcomes in Pediatric Adenotonsillectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Behice Ekici, Associate Professor, PhD, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/05-15
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Adenotonsillar Hypertrophy
Keywords: Adenotonsillectomy; Child; Diet Education; Tonsillectomy Diet; Postoperative Bleeding; Postoperative Pain
MeSH Terms: conditions — Postoperative Hemorrhage; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Parallel Assignment research and control group
Masking Description: research and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- research group (Experimental): The children in the research group and their caregivers will be trained in line with the content of the "Training manual" using lecture and power point presentation methods. Power point presentation training will be given via computer. Before the training, the researcher will briefly introduce himself/herself with a sincere tone of voice to create a reassuring environment. The researcher will then explain the purpose, topic and duration of the study. The researcher will explain to the children and their caregivers that they can express their thoughts or ask questions about the topic during the training
  Interventions: Other: Assigned Interventions (diet training)
- control group (No Intervention): Children in the control group will receive a normal education in line with the clinic functioning. No training on tonsillectomy diet will be given by the investigator.

INTERVENTIONS:
Other: Assigned Interventions (diet training) — Pain and bleeding will be evaluated at 4 hours, 8 hours, 24 hours and 7 days after adenotonsillectomy by using "Wong-Baker Faces Pain Rating Scale" and "Follow-up and Evaluation Form for Children After Adenotonsillectomy in Children".
  Arms: research group

SUMMARY:
This randomized controlled trial aims to evaluate the effect of tonsillectomy diet education on postoperative bleeding and pain in children undergoing adenotonsillectomy. Seventy-six pediatric patients will be randomly assigned to either an intervention group, which will receive specific diet education prior to surgery, or a control group receiving standard care. Bleeding and pain will be assessed at 4, 8, and 24 hours, and on the 7th day after surgery using a specialized follow-up form and the Wong-Baker Faces Pain Rating Scale. The study hypothesizes that diet education will reduce postoperative bleeding and pain, improving recovery and quality of life in children.

DETAILED DESCRIPTION:
Problem Adenotonsillectomy, which means removal of adenoids and tonsils, is one of the most common surgical operations performed in children.The most common indications for tonsillectomy are sleep-disordered breathing, recurrent upper respiratory tract infections, sinusitis, tonsillitis and peritonsillar abscess. Nausea and vomiting, restricted oral intake, high fever, swallowing problems, bleeding and pain are common problems after adenotonsillectomy. Bleeding and pain in the tonsil bed especially after adenotonsillectomy negatively affect the healing process. It leads to a decrease in fluid and food intake and pain control may become difficult. Pain after adenotonsillectomy surgery is a complication that reduces quality of life and may require hospitalization. Pain decreases the quality of life of the child and caregivers after surgery, and children face the risk of decreased oral intake, dehydration due to lack of nutrition and hyperthermia. Another important problem after adenotonsillectomy is bleeding. Postoperative bleeding is one of the most common and serious complications.Bleeding complication may occur in the early or late period. Bleeding within the first 24 hours is classified as primary bleeding, while bleeding that occurs later is called secondary bleeding.It is suggested that primary bleeding is related to acute vascular injuries that occur during surgery, while secondary bleeding is related to fibrinolysis, which can be seen due to clot dissolution in previously coagulated foci as a result of various causes and surgical wound infection. Postoperative bleeding is graded as mild to moderate to severe bleeding according to findings indicating bleeding color and content such as pink, light red with clots, dark red without clots, dark red with clots, ground brown without clots, ground brown with clots in the incision area.A bleeding complication can lead to readmission to hospital after discharge from hospital. Patients admitted with bleeding complications may initially be followed up only with close clinical observation, but in more severe cases, they may require surgical intervention under local or general anesthesia due to bleeding.In addition, bleeding after adenotonsillectomy may rarely result in mortality. Bleeding is more common after adenotonsillectomy surgery as a result of non-compliance with the tonsillectomy diet and consumption of solid, hot, bitter and sour foods. In uncontrolled cases, it is known to cause bleeding that requires a second surgical operation and even fatal bleeding in more advanced cases. In this case, there are precautions to be taken before the complication occurs. These measures are the tonsillectomy diet that should be considered after adenotonsillectomy surgery. It is known that post-adenotonsillectomy bleeding causes psychological social distress and burden on the patient, the patient's relatives and the physician, as well as economic burden.

Method Research Model In this study, the effect of tonsillectomy diet training on bleeding and pain after adenotonsillectomy in children will be examined with a randomized controlled repeated measures design.

Population and Sample The population of the study will consist of children who underwent adenotonsillectomy surgery in the otolaryngology clinic of a public education and research hospital in a district of Istanbul between March and September 2025. In this study, a power analysis was conducted to determine the sample size. Power analysis was performed with G*Power 3.1.9.4 package program.The sample size of the study was calculated with reference to the study of M. Albeladi,2020 due to its similarity to the subject and method of this study, and as a result of the calculations, the effect size was calculated to be 0.95. Accordingly, for the two-tailed hypothesis to maximize the sample size; margin of error α: 0.28 effect size (∆:0.3 and Power: 0.95, the minimum number of children to be included in the study will be 38 children for each group, totaling 76 children.

Training Materials Content of the training manual (I Heal with Cold and Soft Foods) : In the study, the effect of tonsillectomy diet on bleeding and pain after adenotonsillectomy in children will be examined. A training manual will be prepared to ensure the compliance of the child or caregiver with the tonsillectomy diet. In the prepared training manual; general information about adenotonsillectomy surgery and its causes will be briefly explained. What the tonsillectomy diet is, what the diet includes and which foods are appropriate to consume after surgery will be explained. It will be explained which foods should be consumed on which day and which foods should be avoided (bitter, spicy, hard foods, etc.) with tonsillectomy diet. Experts will be consulted to determine the suitability of the content of the training manual to the developmental levels of children and the literature.

Training Power point presentation: Children in the research group and their caregivers will be trained in line with the content of the "Training manual" by using lecture and power point presentation methods. Power point presentation training will be given via computer. Before the training, the researcher will briefly introduce himself/herself in a sincere tone of voice to create a reassuring environment. Then he/she will explain the purpose, subject and duration of the research. The researcher will explain to the children and their caregivers that they can express their thoughts or ask questions about the subject during the training. The routine tonsillectomy diet training given routinely by the clinic nurse will be continued for the children and their caregivers in the control group.

Data and Collection The procedure for data collection will be as follows. Informing the hospital management and health team members: The researcher will have a face-to-face meeting with the hospital administration. In this meeting, information about the research will be given and a date will be determined for obtaining their consent, obtaining ethics committee permission and implementing the research. Data will be collected within the determined date range.

Identification of participant children: Among the children admitted to the otorhinolaryngology clinic for adenotonsillectomy surgery, those who meet the inclusion criteria will be randomly selected by simple randomization.

Obtaining Informed Consents: An "informed consent form" will be obtained from the child and caregiver who accept the study. With the consent to participate in the study, the scope and purpose of the study will be explained in detail to the volunteer family.

Determining the Place, Date and Time of the Training: The training will be held in the room defined for the patient in the inpatient clinic of the otorhinolaryngology clinic in order to facilitate the participation of the children in the research group and their caregivers and to provide a comfortable and quiet environment in the preoperative period. The date and time of the training will be determined one day before the surgery for the children in the study group. The training will be done with direct narration and video animation through the training manual and its duration will be determined as thirty minutes.

Assessment of Bleeding and Pain Pain and bleeding will be evaluated at 4 hours, 8 hours, 24 hours and 7 days after adenotonsillectomy by using "Wong-Baker Faces Pain Rating Scale" and "Follow-up and Evaluation Form for Children After Adenotonsillectomy in Children".

The "Follow-up and Evaluation Form for Children After Adenotonsillectomy" will be evaluated simultaneously by the researcher and the physician in the ward following the child. While pain assessment will be evaluated separately by the 1st (researcher) and 2nd (ward physician) evaluators, bleeding findings will be evaluated and recorded together by the researcher and ward physician. At the beginning of the evaluation form, the month of the evaluation, the reason for the children's admission to the hospital and the average duration of the operation will be evaluated. In this form, the left column includes the color and content of the bleeding. In the 4 columns on the right, the time and number of evaluations of bleeding and pain will be evaluated as 4th hour after surgery 1st evaluation, 8th hour after surgery 2nd evaluation, 24th hour after surgery 3rd evaluation, 7th day after surgery 4th evaluation. The first 3 evaluations will be during hospitalization. The next 7th day evaluation will be evaluated on the 7th day when the child and caregiver are discharged and come for follow-up. The color and content of the bleeding will be evaluated as (pink / clotless, light red / clotless, light red / clotted, dark red / clotless, dark red / clotted, ground brown / clotless, ground brown / clotted). The number of bleeding will be marked as no bleeding, 1 time, 2 times, 3 times or more.

Data Analysis and Interpretation The licensed SPSS (Statistical Package fort he Social Science) 25 package program will be used to evaluate the data. General evaluation of the data and necessary comparisons will be made. During the statistical analysis of the data, the scores obtained from the post-adenotonsillectomy follow-up and evaluation form will be compared as a result of the effect of tonsillectomy diet education on bleeding and pain after adenotonsillectomy surgery, taking into account the age, gender, educational status, previous surgical experiences, age and educational status of the caregiver. Percentage (%) values will be used and statistical analysis methods will be used to examine whether there are significant differences between these data. Descriptive statistical methods (number, percentage, mean, standard deviation, median) as well as Shapiro-Wilks test will be used to evaluate the normal distribution. Independent t-test will be used to compare paired groups.

ELIGIBILITY:
Inclusion Criteria:

* The child being sick,
* The child will have an adenotonsillectomy,
* The child has no milk allergy (to exclude children at risk of developing milk allergy during the data collection process),
* The child's caregiver stays with the child during the research process (to avoid communication barriers and disruptions in treatment and care instructions during the training and data collection process),
* The child and caregiver can speak and understand Turkish (to avoid communication barriers during the training and data collection process),
* The child's caregiver agrees to the research,
* Children without swallowing difficulties and aspiration risk (e.g. nasogastric catheter, tracheostomy)
* Children without diseases that cause maladaptive behavior (e.g. autism, cerebral palsy)

Exclusion Criteria:

* The child has a milk allergy,
* Children with diseases that cause swallowing difficulties, risk of aspiration and maladaptive behavior (e.g. autism, cerebral palsy)
* Failure of the child and caregiver to attend the follow-up examination on the 7th day after surgery

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Follow-up and Evaluation Form for Children After Adenotonsillectomy | 4th hour after surgery 1st assessment, 8th hour after surgery 2nd assessment, 24th hour after surgery 3rd assessment, 7th day after surgery 4th assessment. The first 3 assessments will be duri
  The time and number of evaluations; 4th hour after surgery will be considered as 1st evaluation, 8th hour after surgery as 2nd evaluation, 24th hour after surgery as 3rd evaluation, 7th day after surgery as 4th evaluation. The first 3 evaluations will be during hospitalization. The next 7th day evaluation will be evaluated on the 7th day when the child and caregiver are discharged and come for follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal AKDENİZ, Principal Investigator — Maltepe University School of Nursing İstanbul, Turkey
Locations (1):
- Hilal AKDENİZ, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Windfuhr JP, Chen YS, Remmert S. Hemorrhage following tonsillectomy and adenoidectomy in 15,218 patients. Otolaryngol Head Neck Surg. 2005 Feb;132(2):281-6. doi: 10.1016/j.otohns.2004.09.007. PMID 15692542
- [Background] Bellis JR, Pirmohamed M, Nunn AJ, Loke YK, De S, Golder S, Kirkham JJ. Dexamethasone and haemorrhage risk in paediatric tonsillectomy: a systematic review and meta-analysis. Br J Anaesth. 2014 Jul;113(1):23-42. doi: 10.1093/bja/aeu152. PMID 24942713
- [Background] Gulsen S, Cikrikci S. Comparison of Endoscope-Assisted Coblation Adenoidectomy to Conventional Curettage Adenoidectomy in Terms of Postoperative Eustachian Tube Function. J Craniofac Surg. 2020 Jun;31(4):919-923. doi: 10.1097/SCS.0000000000006039. PMID 31764564
- [Background] Meybodian M, Dadgarnia M, Baradaranfar M, Vaziribozorg S, Mansourimanesh M, Mandegari M, Saeidi Eslami N. Effect of Cold Diet and Diet at Room Temperature on Post-Tonsillectomy Pain in Children. Iran J Otorhinolaryngol. 2019 Mar;31(103):81-86. PMID 30989073
- [Background] Ashbach MN, Ostrower ST, Parikh SR. Tonsillectomy techniques and pain: a review of randomized controlled trials and call for standardization. ORL J Otorhinolaryngol Relat Spec. 2007;69(6):364-70. doi: 10.1159/000108369. Epub 2007 Nov 23. PMID 18033974
- [Background] Boroumand P, Zamani MM, Saeedi M, Rouhbakhshfar O, Hosseini Motlagh SR, Aarabi Moghaddam F. Post tonsillectomy pain: can honey reduce the analgesic requirements? Anesth Pain Med. 2013 Summer;3(1):198-202. doi: 10.5812/aapm.9246. Epub 2013 Jul 1. PMID 24223362
- [Background] Ostvoll E, Sunnergren O, Ericsson E, Hemlin C, Hultcrantz E, Odhagen E, Stalfors J. Mortality after tonsil surgery, a population study, covering eight years and 82,527 operations in Sweden. Eur Arch Otorhinolaryngol. 2015 Mar;272(3):737-43. doi: 10.1007/s00405-014-3312-z. Epub 2014 Oct 2. PMID 25274044
- [Background] Brasher C, Gafsous B, Dugue S, Thiollier A, Kinderf J, Nivoche Y, Grace R, Dahmani S. Postoperative pain management in children and infants: an update. Paediatr Drugs. 2014 Apr;16(2):129-40. doi: 10.1007/s40272-013-0062-0. PMID 24407716
- [Background] Albeladi MA, Salamah MA, Alhussaini R. The Effect of Ice Cream Intake on Pain Relief for Patients After Tonsillectomy. Cureus. 2020 Jul 9;12(7):e9092. doi: 10.7759/cureus.9092. PMID 32789040
- [Background] Soleymanifard F, Khademolhoseyni SM, Nouri JM. Nursing process in post tonsillectomy pain diagnosis: a systematic review. Glob J Health Sci. 2014 Aug 22;7(1):180-7. doi: 10.5539/gjhs.v7n1p180. PMID 25560345
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343